CLINICAL TRIAL: NCT00904709
Title: The Assessment of the Minimal Effective and Tolerated Dose of Tranexamic Acid in Women With Menorrhagia Who Have Bleeding Disorders
Brief Title: The Assessment of Tranexamic Acid in Women With Menorrhagia Who Have Bleeding Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: K. Sue Robinson (Other)
Collaborators: Canadian Hemophilia Society (Other)
Responsible Party: Sponsor-Investigator, K. Sue Robinson, hematologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RS/2009-341
Record Dates: First submitted 2009-05-15; First posted 2009-05-20 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Menorrhagia
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tranexamic acid, Menorrhagia, Bleeding (Experimental): Tranexamic acid with titrated doses. All women with menorrhagia will take .
  Interventions: Drug: tranexamic acid

INTERVENTIONS:
Drug: tranexamic acid — After The starting dose of tranexamic acid will be 500 mg twice daily beginning the first day of menstrual flow for a total of 6 days per menstrual cycle. If after 2 days there is still menorrhagia without significant side effects the will be increased. The women will be assessed again at day 4 and 9 and dose escalation will continue until they have reached the optimal dose.The dose of tranexamic acid will be increased as follows: 1000 mg twice daily, 1000 mg three times daily, 1500 mg/1000 mg/1000 mg, 1000 mg four times daily, 1500 mg three times daily, and 1500 mg four times daily (maximum dose).Each patient will be followed for a minimum of one menstrual cycle and a maximum of 3 cycles.
  Other Names: Cyklokapron

SUMMARY:
Many women have heavy periods and this can be associated with low blood, tiredness and inability to carry out normal activities. Approximately 10-30% of these women will have an underlying bleeding disorder. There is a drug called tranexamic acid which is commonly used and is effective in reducing menstrual flow. However, up to 1/3 of women have side effects and they are more common at higher doses. In the medical literature, there are different dosing schedules and there is one commonly recommended in Canada. Women with underlying bleeding disorders may require higher doses of this medication compared to those who do not. In this study, the investigators want to find the lowest effective dose of tranexamic acid for girls and women with heavy periods who have bleeding disorders and the investigators think this will be lower then the usual recommended dose. If the investigators' results support this, it may contribute to changing how the investigators presently prescribe this medication and may provide a better option for women with heavy periods in particular those with bleeding disorders. The investigators have just started a Women with Bleeding Disorders Clinic and hope that this project will lead to better care for the patients and more research in the future.

DETAILED DESCRIPTION:
Menorrhagia, or heavy menstrual bleeding, represents an important health issue for premenopausal women and is a common cause for primary care consultations. Approximately 10-15% of women have heavy periods. This may be associated with iron deficiency anemia, fatigue, and time lost from school, work and regular activities. Up to 50% of women with menorrhagia who have an underlying bleeding disorder have functional limitations and reduction of quality of life during their menstrual period.

The literature reports that 10-30% of women with menorrhagia have an underlying bleeding disorder. The American Society of Hematology highlighted this as a major public health issue in 2006, and there have been ongoing efforts to address this problem. The prevalence of a bleeding disorder in the normal population is 1 in 100; von Willebrand Disease (VWD) being the most common. Studies have shown between 57% and 93% of women with bleeding disorders have menorrhagia. Therefore, women, who present with menorrhagia, should be considered for investigation of a bleeding disorder.

Obtaining an accurate history of menorrhagia from women is often difficult for several reasons. Women may be reluctant to initiate discussion about their heavy periods. Also, women with underlying hereditary bleeding disorders may have heavy periods but since they are the same as other affected women in their families they consider their menses "normal." Not infrequently,a mild bleeding disorder may go undiagnosed until adulthood.

Menorrhagia is objectively defined as menstrual blood loss of > 80mls. It is well known that assessment of menstrual blood loss by history alone is unreliable and inaccurate. The alkaline hematin method provides an objective and accurate technique for the measurement of menstrual blood loss and is considered the gold standard. However this method is time-consuming, not readily available for clinical use and impractical, as it requires women to collect all of their sanitary products for an entire menstrual cycle. The pictorial blood assessment chart (PBAC) is a simple, non-laboratory method that provides a semi-quantitative assessment of menstrual flow. Using this method, the patient records the number and degree of saturation of pads and/or tampons used for up to 8 days of their menstrual cycle on a pictorial chart and a corresponding score is calculated. In their original report, Higham et al defined menorrhagia as a PBAC score of > 100 with a sensitivity of 86% and a specificity of 81 %. Janssen et al later reported that a cut-off score of 185 provides high positive and negative predictive values for 'true' menorrhagia as opposed to the score of > 100 that was not validated by Reid et al, in a more recent publication. In both the Higham and the Janssen studies the confidence intervals of the estimates of sensitivity were not reported, therefore it is difficult to select either one as being definitively better to use as a cut-off score. In our study we have decided to use a cut-off PBAC score of 100 as a more conservative approach that will allow the inclusion of more patients with heavy menstrual flow.

There are a number of treatment options for women with menorrhagia including hormone therapy (combined oral estrogen/progesterone, progesterone alone), tranexamic acid (and other antifibrinolytic agents), danazol, non steroidal anti-inflammatory drugs (NSAIDs), progesterone releasing intrauterine devices, and, finally, the surgical options of endometrial ablation and hysterectomy. An additional therapy, for women with certain bleeding disorders (VWD, platelet dysfunction and Hemophilia A carriers) is desmopressin (DDAVP) (intranasal or subcutaneous). Tranexamic acid is a first line therapy for women with menorrhagia who do not require contraception and who prefer non-hormonal therapy. It is considered standard therapy around the world and in most countries (e.g. Canada), it is available by prescription only, but interestingly in Sweden it is obtained 'over-the-counter.'

Antifibrinolytic therapy has been used for almost forty years for menorrhagia - the first publication was in 1965. It has previously been described that fibrinolysis is increased in the menstrual fluid and endometrium in women with heavy menstrual flow. Tranexamic acid, which is a fibrinolytic inhibitor, competitively blocks the activation of plasminogen to plasmin and thereby reducing fibrinolysis. Tranexamic acid reduces menstrual blood loss by up to 50% and it has been shown to be at least as equally as effective as oral contraceptives, NSAIDs, and intranasal desmopressin. There is no consensus as to the minimal effective dose, the dose scheduling and the optimal duration of therapy. In the published literature, the effective dose is variable and ranges from 1000 mg/day to 6000 mg/day. The recommended dose by the Compendium of Pharmaceuticals and Specialties (CPS), 2009, published by the Canadian Pharmacists Association, is 3000 mg/day to 6000 mg/day. The current recommended dose as per the Clinical Practice Guidelines for the Management of Abnormal Uterine Bleeding by the Society of Obstetricians and Gynecologists of Canada and the Canadian Hemophilia Society document on the Management of Women with Bleeding Disorders is 1000 mg orally four times a day. Interestingly, in China, it is recommended to give 2000 mg/day. The recommended duration of therapy is also variable; the CPS states the medication should be started "when the flow is copious" and taken for "several days." Most clinical trials have used a 4-5 day duration of therapy. It is given in different schedules, most commonly 3 to 4 times per day. A recent study compared two doses of tranexamic acid, 2000 mg/day vs. 1000 mg/day, both doses given on a twice-a-day schedule, with an additional placebo arm, assessing the effect on prevention of menorrhagia in women with intrauterine devices (IUDs). The women randomized to the tranexamic acid arms had significantly less menstrual flow compared with the placebo group and there was no significant difference in efficacy between the two doses of tranexamic acid. Women with underlying bleeding disorders may need higher doses than women without bleeding disorders; however, this is uncertain. This medication is not without toxicity and up to one-third of women experience side effects that are dose dependant. The most common adverse effects are nausea, vomiting, diarrhea and, less common, are headaches, dizziness and allergic reaction. Tranexamic acid is expensive; the retail price is $1.34/500-mg capsule. For example a dose of 4000 mg/day for 5 days would cost a patient $64.34/month including the dispensing fee. Common reasons for discontinuing the medication include side effects, cost and the inconvenience associated with multiple dosing. Many patients will adjust their dose - finding a balance of efficacy, minimal toxicity, cost, and frequency of dosing. It is our experience that some patients find this balance with a minimal dose of 500 mg taken twice daily. In this study we propose to investigate whether the minimal effective and tolerated dose of tranexamic acid, based on the PBAC score, quality of life factors, and tolerability of side effects is less than the current Canadian recommended dose of 1000 mg orally four times a day.

Study Objectives:

* Primary Objective

  * To determine if the minimal effective and tolerated dose of tranexamic acid for girls and women with menorrhagia who have bleeding disorders is lower than the current dose of 1000 mg orally, four times a day, as recommended by the Clinical Practice Guidelines for the Management of Abnormal Uterine Bleeding by the Society of Obstetricians and Gynecologists of Canada and the Canadian Hemophilia Society document on the Management of Women with Bleeding Disorders.
* Secondary Objectives

  * To determine an accurate estimate of the proportion of women who present to our clinics with menorrhagia who have an underlying bleeding disorder. Based on the literature this is expected to be 10%-30%.
  * To determine the effect of body mass index (BMI), age, dose-related side effects, concurrent medications and quality of life factors on the optimal dose of tranexamic acid.

Study hypotheses:

* Primary hypothesis

  * The minimal effective and tolerated dose of tranexamic acid required by women with menorrhagia who have bleeding disorders is lower than the current Canadian recommendation of 1000 mg orally, four times daily (4000 mg/day).
* Secondary hypotheses

  * The true proportion of women with menorrhagia who have bleeding disorders is under-reported.
  * Women with menorrhagia without bleeding disorders require a lower dose of tranexamic acid than women with menorrhagia with bleeding disorders.
  * In addition to the presence of a bleeding disorder, there are likely other factors including age, BMI, tolerance of side effects, subjective assessment of bleeding, quality of life issues and compliance that impact on the dosing of tranexamic acid in women with menorrhagia.
  * A decision tool can be developed to aid in dosing women with menorrhagia based on risk factors such as the presence of a bleeding disorder, age and BMI.

ELIGIBILITY:
Inclusion Criteria:Clinical diagnosis of Menorrhagia

* Must be able to swallow tablets

Exclusion Criteria:

* Endometrial abnormality
* Pelvic infection
* Pregnancy
* Breast Feeding
* Requirement for birth control
* Known intolerance/lack of effect of tranexamic acid

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 249 (Actual)
Dates: Start 2009-10-19 (Actual); Primary Completion 2014-03-01 (Actual); Study Completion 2014-03-01 (Actual)

PRIMARY OUTCOMES:
Minimal effective dose of tranexamic acid | 4 months

SECONDARY OUTCOMES:
Quality of Life Assessment | 4 months